CLINICAL TRIAL: NCT02613767
Title: Muscle Protein Synthesis Rates After Protein Consumption in Lean, Overweight, and Obese Adults
Status: Completed | Type: Observational
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Principal Investigator, Nicholas Burd, Assistant Professor, University of Illinois at Urbana-Champaign
Other Study IDs: 15161
Record Dates: First submitted 2015-11-05; First posted 2015-11-24 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — guar meal protein, Cyamopsis tetragonoloba

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples and Skeletal muscle tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Obese: BMI >30 kg/m2, Protein meal,
  L-[ring 13C6]Phenylalanine infusion
  Interventions: Other: Protein meal; Other: L-[ring 13C6]Phenylalanine infusion
- Overweight: BMI >25 and < 30 kg/m2, Protein meal,
  L-[ring 13C6]Phenylalanine infusion
  Interventions: Other: Protein meal; Other: L-[ring 13C6]Phenylalanine infusion
- Healthy-Weight: BMI >18 and < 25 kg/m2, Protein meal,
  L-[ring 13C6]Phenylalanine infusion
  Interventions: Other: Protein meal; Other: L-[ring 13C6]Phenylalanine infusion

INTERVENTIONS:
Other: Protein meal — Ingestion of protein
Other: L-[ring 13C6]Phenylalanine infusion — experimental method for determining protein synthesis rates

SUMMARY:
There are an increasing number of individuals in the United States with obesity, and this is a major health concern with links to many chronic diseases. Impairments in protein metabolism with obesity may disrupt muscle function and modify the dietary protein requirements in obese individuals. Further, overweight and obese type 2 diabetics exhibit dramatically reduced skeletal muscle mass compared with lean, healthy controls. Surprisingly, the influence of being overweight or obese on this decline in muscle mass remains understudied, despite clear evidence that similar metabolic impairments typically exist in these populations prior to the development of overt diabetes. Protein ingestion provides the amino acid building blocks to synthesize and repair muscle proteins in adults. Previous research has shown that the muscle protein synthetic response to food ingestion may be reduced in overweight/obese adults. However, this research provided the 'free' amino acids in small portions every 15 min during the postprandial period. In free living conditions, however, it is more common to consume protein dense foods in single portions. Currently, there is no information available on how eating protein rich foods affects muscle protein synthesis in overweight and obese adults. This proposed research will fill this research gap by being the first study to compare the muscle protein synthetic response to the ingestion of a meal-like amount of high quality protein in lean, overweight and obese adults. The objective of this study is to determine the muscle protein synthetic response after the consumption of 35g pork protein in lean, overweight and obese adults. In order to assess this objective the researchers propose to use primed continuous infusion of L-[ring-13C6] phenylalanine to measure muscle protein synthesis rates after the consumption of dietary protein. In a parallel design the researchers will study 13 obese (BMI 30-39.9 kg/m2) participants, 13 overweight (BMI 25-29.9 kg/m2), and 13 age-matched lean controls (BMI 18-24.9 kg/m2) between the ages of 20 and 45 years. All subjects will be sedentary and weight stable for the previous 6 months. On the test day, subjects will remain sedentary for the determination of muscle protein synthesis in both the fasted state and after consumption of the protein meal. Blood and muscle sampling will occur on the test day.

DETAILED DESCRIPTION:
Participants will be asked to report to the laboratory at 7:00 am following an overnight fast. Upon arrival, a Teflon catheter will be inserted in an antecubital vein of one arm for arterialized blood sampling and a baseline blood sample will be drawn. Arterialized blood samples will be obtained by wrapping the subjects' forearm in a heating blanket (45 °C) for 10 min prior to each blood collection time point. A second Teflon catheter will be inserted in an antecubital vein of the opposite arm, and participants will receive a priming dose of L-[ring- 13C6]phenylalanine (2.0 µmol∙kg) prior to initiating a continuous infusion of L-[ring-13C6]phenylalanine (0.05 µmol∙kg∙min) (t=-240). The prime and continuous tracer infusion will be passed through a 0.2 μm filter. Blood will be collected every 1 hour and biopsies of the vastus lateralis will be collected at t=-180 and t=-15 min using a 5 mm Bergström needle (modified for manual suction) under 2% xylocaine local anesthesia for the measurement of postabsorptive muscle protein synthesis rates. The second biopsy (t=-15 min) will be used to determine baseline levels of phosphorylated and total proteins involved in nutrient sensing and muscle anabolic signaling. Subsequently, the participants will ingest 6 oz of fresh ground center cut pork loin. This cut of meat was selected due to its low lipid content (2.5-3%) and it is uniform in shape, size and composition. Along with the ingested pork, the participants will consume 300 mL of water. The water will be enriched to 5% with tracer according to the phenylalanine content of ~4% in the pork. This approach is required to minimize disturbances in isotopic steady state and provide appropriate conditions for the calculation of postprandial muscle protein synthesis rates. The time required to consume the pork will be recorded. The completion of the pork meal and water will mark the start of the postprandial phase (t=0). During this period, arterialized blood samples will be collected into evacuated chilled heparinized tubes at t=30, 60, 90, 120, 180, 240, and 300 min. Additional muscle biopsies will be collected at t=120 and 300 min of the experimental infusion for the measurement of postprandial muscle protein synthetic and muscle anabolic signaling protein responses. The muscle biopsy samples will be freed from any visible blood, fat, and connective tissue, rapidly frozen in liquid nitrogen and stored at -80˚C until analysis. Blood samples will be centrifuged at 1,000×g at 4˚C for 10 min and separated plasma will be transferred to 2.0 ml cryovials. The plasma samples will be stored at -20˚C until further analysis.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females
* Aged between 20-45 years
* Healthy, sedentary
* Three groups, age and sex matched
* Healthy weight group: BMI 18-24.9 kg/m2
* Overweight group: BMI 25-29.9 kg/m2
* Obese group: BMI 30-39.9 kg/m2

Exclusion Criteria:

* Smoking
* Allergies to pork consumption
* Unusually high protein consumption
* Vegetarians
* Phenylketonuria (PKU)
* Diagnosed GI tract diseases
* Arthritic conditions
* A history of neuromuscular problems
* Previous participation in amino acid tracer studies
* Predisposition to hypertrophic scarring or keloid formation
* Individuals on any medications known to affect protein metabolism (i.e. corticosteroids, non-steroidal anti-inflammatories, or prescription strength acne medications).
* Irregular menstrual cycles during the previous year
* Pregnancy
* High BMI that is not representative of being overweight or obese (e.g. resistance trained individuals, football players)

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: We recruited 32 healthy, sedentary adult subjects (20-45 y) for this investigation. There are three groups being studied, which will be stratified by body mass index. Because randomization is not possible, groups were balanced by age and sex. No races or ethnic groups will be specifically recruited or excluded.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2014-12; Primary Completion 2015-09 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Fractional synthetic rate of myofibrillar proteins | 7 hours

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas A Burd, Ph.D, Principal Investigator — Assistant Professor

REFERENCES:
- [Derived] Beals JW, Mackenzie RWA, van Vliet S, Skinner SK, Pagni BA, Niemiro GM, Ulanov AV, Li Z, Dilger AC, Paluska SA, De Lisio M, Burd NA. Protein-Rich Food Ingestion Stimulates Mitochondrial Protein Synthesis in Sedentary Young Adults of Different BMIs. J Clin Endocrinol Metab. 2017 Sep 1;102(9):3415-3424. doi: 10.1210/jc.2017-00360. PMID 28911136
- [Derived] Beals JW, Sukiennik RA, Nallabelli J, Emmons RS, van Vliet S, Young JR, Ulanov AV, Li Z, Paluska SA, De Lisio M, Burd NA. Anabolic sensitivity of postprandial muscle protein synthesis to the ingestion of a protein-dense food is reduced in overweight and obese young adults. Am J Clin Nutr. 2016 Oct;104(4):1014-1022. doi: 10.3945/ajcn.116.130385. Epub 2016 Sep 7. PMID 27604771